CLINICAL TRIAL: NCT01999647
Title: Intraneural Injection of Ropivacaine for Subgluteal Sciatic Nerve Block Leads to Faster Onset and Higher Success Rates: a Randomized, Controlled Trial
Brief Title: Efficacy of Ultrasound-Guided Local Anesthetic Injection Into or Around the Sciatic Nerve for Lower Limb Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Marco Baciarello, Assistant Professor of Anesthesiology, Critical Care and Pain Medicine, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANEST-ORT-04
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Orthopedic Disorders; Foot Diseases; Injuries, Leg; Injuries, Foot; Injuries, Knee
Keywords: Lower Extremity; Sciatic Nerve; Anesthetics, Local; Ropivacaine; Ultrasonography
MeSH Terms: conditions — Musculoskeletal Diseases; Foot Diseases; Leg Injuries; Foot Injuries; Knee Injuries | interventions — Passive Cutaneous Anaphylaxis; Ropivacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineural (Active Comparator): Patients in this group will receive a perineural injection for subgluteal sciatic nerve block under real-time, short-axis, in-plane ultrasound guidance, in addition to a femoral nerve block and patient-controlled postoperative analgesia. Ropivacaine will be used for the sciatic nerve block, whereas the choice of agent for the femoral nerve block is left to the attending anesthesiologist.
  Interventions: Procedure: Perineural Injection for Subgluteal Sciatic Nerve Block; Procedure: Femoral Nerve Block; Procedure: Patient-Controlled Postoperative Analgesia; Drug: Ropivacaine
- Intraneural (Experimental): Patients in this group will receive an intraneural injection for subgluteal sciatic nerve block under real-time, short-axis, in-plane ultrasound guidance, in addition to a femoral nerve block and patient-controlled postoperative analgesia. Ropivacaine will be used for the sciatic nerve block, whereas the choice of agent for the femoral nerve block is left to the attending anesthesiologist.
  Interventions: Procedure: Intraneural Injection for Subgluteal Sciatic Nerve Block; Procedure: Femoral Nerve Block; Procedure: Patient-Controlled Postoperative Analgesia; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Intraneural Injection for Subgluteal Sciatic Nerve Block — The injection will start as the needle penetrates the outermost discernible layer of the nerve (epineurium) under ultrasound guidance. The injection will be adjudicated as "intraneural" if nerve cross section expansion and a reduction in echogenicity are observed.
  Short-axis real-time ultrasound imaging will be used, with an in-plane needle approach.
  Other Names: Injection beneath the common investing extraneural layer; Subepineural Injection; Gluteal sciatic nerve block; Subparaneural injection
  Arms: Intraneural
Procedure: Perineural Injection for Subgluteal Sciatic Nerve Block — The injection will start as the needle indents the outermost discernible layer of the nerve (epineurium) under ultrasound guidance. The injection will be adjudicated as "intraneural" if the drug infiltrates the space between the epimysium of the surrounding muscles and the outer epineurium of the sciatic nerve.
  Short-axis real-time ultrasound imaging will be used, with an in-plane needle approach.
  Other Names: Injection outside the common investing extraneural layer; Epineural injection; Extraneural injection; Injection outside the paraneurium
  Arms: Perineural
Procedure: Femoral Nerve Block — Patients will receive an ultrasound-guided femoral nerve block using a short- or long-acting local anesthetic, as deemed indicated.
Procedure: Patient-Controlled Postoperative Analgesia — Patients will receive a patient-controlled intravenous or perineural catheter-based analgesia, depending on their preference and the anesthesiologist's indication.
  Other Names: PCA; PCIVA; PCCPNB; Patient-controlled continuous peripheral nerve block
Drug: Ropivacaine — Thirty milliliters of 0.75% (wt/vol) ropivacaine will be used for the sciatic nerve block.
  Other Names: Local Anesthetic; Naropin; Naropine

SUMMARY:
This study was designed to assess whether the injection of local anesthetic into the nerve (intraneural), as opposed to around it (perineural), requires a shorter time to develop surgical anesthesia of the lower leg.

The investigators will compare the two types of injection using the same drug, so as to determine if there is an actual difference onset time. They will also examine the overall success rate of either kind of sciatic nerve blocks as the sole anesthetic for non-emergent orthopedic surgery.

The safety of these procedures will be examined by in-hospital and phone-call follow-up contacts.

DETAILED DESCRIPTION:
This will be a randomized, controlled, patient- and observer-blinded trial assessing block characteristics after intra- or perineural injection of ropivacaine for subgluteal sciatic nerve blocks performed for elective surgery of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non-emergent orthopedic procedure of knee, leg, foot with thigh tourniquet
* ASA Physical Status Class I-III
* Consenting to surgery under peripheral nerve block anesthesia (sciatic + femoral/saphenous block)

Exclusion Criteria:

* Unable to understand or communicate for the purpose of the study
* Exhibiting any neurological disturbance of the ipsilateral lower extremity
* Inability to satisfactorily image the sciatic nerve in the opinion of the attending anesthesiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Onset Time of Sciatic Nerve Block | ≤30 minutes after block performance
  Time to onset of sciatic nerve anesthesia, defined as both following criteria:
  * Sensory: does not feel pain or discomfort when pricked with a 25G needle.
  * Motor: able to slightly curl toes; unable to flex the ankle.

SECONDARY OUTCOMES:
Success Rate of Sciatic Nerve Blocks | ≤30 min after block performance
  The percentage of patients who attain the criteria for block success within 30 minutes of the injection.
  Investigators will also report the percentage of patients who successfully complete surgery without significant additional analgesia (see below); this will be defined as "clinical success rate."
Incidence and Prevalence of Neurologic Disturbances | 30 days after anesthesia performance
  Patients will be interviewed at ~4 h (block resolution visit), 7 days and (if necessary) at 30 days to assess for residual neurologic disturbances in the sciatic nerve territory.
  The incidence/prevalence of these phenomena will be noted.
Differences in Time to Resolution of Sciatic Nerve Block | <12 h
  The time at which sensory and motor function of the sciatic nerve have recovered at least to the following criteria:
  * Sensory: patients feel discomfort when pricked with a thin needle (25G)
  * Motor: patients may move both toes and ankle, albeit with reduced strength
  This outcome measure will be examined by an investigator every 30-60 min and reported by patients as "time to return of sensation and movement". The investigator-reported value will be preferred if both are available.

OTHER OUTCOMES:
Extra- vs. Intraneural Minimum Electrical Stimulation Thresholds | During performance of nerve block (<30 min)
  The minimum electrical nerve stimulation threshold will be recorded as a function of needle tip position.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Baciarello, MD, Principal Investigator — University of Parma
Locations (1):
- Anesthesia, Critical Care and Pain Medicine - University of Parma, Parma, PR, Italy

REFERENCES:
- [Background] Tran DQ, Dugani S, Pham K, Al-Shaafi A, Finlayson RJ. A randomized comparison between subepineural and conventional ultrasound-guided popliteal sciatic nerve block. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):548-52. doi: 10.1097/AAP.0b013e318235f566. PMID 22005661
- [Background] Andersen HL, Andersen SL, Tranum-Jensen J. Injection inside the paraneural sheath of the sciatic nerve: direct comparison among ultrasound imaging, macroscopic anatomy, and histologic analysis. Reg Anesth Pain Med. 2012 Jul-Aug;37(4):410-4. doi: 10.1097/AAP.0b013e31825145f3. PMID 22609646
- [Background] Robards C, Hadzic A, Somasundaram L, Iwata T, Gadsden J, Xu D, Sala-Blanch X. Intraneural injection with low-current stimulation during popliteal sciatic nerve block. Anesth Analg. 2009 Aug;109(2):673-7. doi: 10.1213/ane.0b013e3181aa2d73. PMID 19608846